CLINICAL TRIAL: NCT01874145
Title: An Open-Label, Randomized, Multi-Center, Parallel-Arm Study to Assess the Safety and Tolerability of Glatiramer Acetate 40 mg/mL Three Times a Week Compared to 20 mg/mL Daily Subcutaneous Injections in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Safety and Tolerability of Glatiramer Acetate
Acronym: GLACIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-MS-303
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Glatiramer Acetate; Glatiramer
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GA 20 mg/mL every day (Active Comparator): Glatiramer acetate (GA) 20 mg in 1 mL SC injection administered every day (QD) for the 4 months of the core study.
  Interventions: Drug: GA 20 mg/mL
- GA 40 mg/mL 3 times a week (Experimental): Glatiramer acetate (GA) 40 mg in 1 mL SC injection administered three times a week (TIW) for the 4 months of the core study.
  During the Extension period, all participants to continue treatment with GA 40 mg/mL TIW until this dose regimen is commercially available for the treatment of RRMS patients.
  Interventions: Drug: GA 40 mg/mL

INTERVENTIONS:
Drug: GA 20 mg/mL — Glatiramer acetate (GA) 20 mg/mL subcutaneous (SC) injection, the commercial product, is a single-use pre-filled syringe (PFS) containing 1.0 ml of a clear, colorless to slightly yellow, sterile, non-pyrogenic solution.
  Other Names: Glatiramer Acetate; Copaxone®
  Arms: GA 20 mg/mL every day
Drug: GA 40 mg/mL — Glatiramer acetate (GA) 40 mg/mL subcutaneous (SC) injection, is a single-use pre-filled syringe (PFS) containing 1.0 ml of a clear, colorless to slightly yellow, sterile, non-pyrogenic solution.
  Other Names: Glatiramer Acetate; Copaxone®
  Arms: GA 40 mg/mL 3 times a week

SUMMARY:
This is an open-label, randomized, multi-center, parallel-arm study to assess the safety and tolerability of a daily dose of Glatiramer Acetate (GA) 40 mg/mL three times a week (TIW) administered subcutaneously (SC) as compared to GA 20 mg/mL every day (QD) administered SC.

DETAILED DESCRIPTION:
The study will comprise of a Core study and an Extension phase. During the Core study, subjects will be evaluated at study sites for 5 scheduled visits at Months: -1 (Screening), 0 (Baseline), 1, 2, and 4 (Termination/Early Termination). Subjects who complete all scheduled visits will have final procedures and assessments performed at the final visit (Month 4, Termination visit). Subjects who withdraw from the study before completing the 4 months evaluation period will have Early Termination (ET) procedures and assessments performed at their final visit.

During the Extension phase, all subjects will be offered to continue treatment with GA 40 mg/mL TIW. Subjects will be evaluated every 4 months until this dose strength is commercially available for the treatment of Relapsing-Remitting Multiple Sclerosis (RRMS) patients or until the development of this GA dose regimen is stopped by the Sponsor, the last visit of this phase will be called Termination/ET-Extension visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years of age or older
2. Subjects must have a confirmed and documented RRMS diagnosis as defined by the Revised McDonald criteria, with relapse onset disease or a relapsing-remitting disease course
3. Subjects must be ambulatory with a Kurtzke Expanded Disability Status Scale (EDSS) score of 0-5.5 in both the Screening and Baseline visits.
4. Subjects must be in a stable neurological condition, relapse-free and free of any corticosteroid treatment [intravenous (IV), intramuscular (IM) and/or per os (PO)] or adrenocorticotrophic hormone (ACTH), 60 days prior to randomization.
5. Subjects must be treated with Glatiramer Acetate (GA) 20mg/mL QD SC injection for a minimum of 6 months prior to screening.
6. Women of child-bearing potential must practice an acceptable method of birth control [acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, oral contraceptives, contraceptive patch, long-acting injectable contraceptive, partner's vasectomy or a double-barrier method (condom or diaphragm with spermicide)].
7. Subjects must be able to sign and date a written informed consent prior to entering the study.
8. Subjects must be willing and able to comply with the protocol requirements for the duration of the study

Exclusion Criteria:

1. Subject has any contraindication to Glatiramer Acetate therapy
2. Subjects with progressive forms of multiple sclerosis (MS).
3. Subjects with Neuromyelitis Optica (NMO).
4. Use of experimental or investigational drugs, and/or participation in drug clinical studies within the 6 months prior to screening.
5. Concomitant use of other disease modifying drug for MS ((Fingolimod (Gilenya®), dimethyl fumarate (Tecfidera®), Teriflunomide (Aubagio®) or intravenous immunoglobulin (IVIG)) within 6 months prior to screening
6. Previous use of mitoxantrone, cladribine, alemtuzumab, rituximab, natalizumab.
7. Chronic (more than 30 consecutive days) systemic (IV, PO or IM) corticosteroid treatment within 6 months prior to screening visit.
8. Previous total body irradiation or total lymphoid irradiation.
9. Previous stem-cell treatment, autologous bone marrow transplantation or allogenic bone marrow transplantation.
10. Pregnancy or breastfeeding.
11. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation, as determined by medical history, physical exams, ECG and abnormal laboratory tests. Such conditions may include hepatic, renal or metabolic diseases, systemic disease, acute infection, current malignancy or recent history (5 years) of malignancy, major psychiatric disorder, history of drug and/or alcohol abuse and allergies that could be detrimental according to the investigator's judgment.
12. Subjects who underwent endovascular treatment for Chronic Cerebrospinal Venous Insufficiency (CCSVI).
13. Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Teva Investigational Site 10706, Cullman, Alabama
  - Teva Investigational Site 10719, Gilbert, Arizona
  - Teva Investigational Site 10720, Phoenix, Arizona
  - Teva Investigational Site 10727, Fresno, California
  - Teva Investigational Site 10731, Long Beach, California
  - Teva Investigational Site 10735, Newport Beach, California
  - Teva Investigational Site 10712, Oceanside, California
  - Teva Investigational Site 10708, Centennial, Colorado
  - Teva Investigational Site 10715, Maitland, Florida
  - Teva Investigational Site 10718, Pompano Beach, Florida
  - Teva Investigational Site 10709, St. Petersburg, Florida
  - Teva Investigational Site 10707, Tampa, Florida
  - Teva Investigational Site 10711, Tampa, Florida
  - Teva Investigational Site 10710, Northbrook, Illinois
  - Teva Investigational Site 10734, Indianapolis, Indiana
  - Teva Investigational Site 10732, Baltimore, Maryland
  - Teva Investigational Site 10726, Great Falls, Montana
  - Teva Investigational Site 10702, Henderson, Nevada
  - Teva Investigational Site 10717, Patchogue, New York
  - Teva Investigational Site 10723, Plainview, New York
  - Teva Investigational Site 10716, Charlotte, North Carolina
  - Teva Investigational Site 10724, Raleigh, North Carolina
  - Teva Investigational Site 10721, Winston-Salem, North Carolina
  - Teva Investigational Site 10733, Bellevue, Ohio
  - Teva Investigational Site 10703, Columbus, Ohio
  - Teva Investigational Site 10714, Dayton, Ohio
  - Teva Investigational Site 10704, Uniontown, Ohio
  - Teva Investigational Site 10725, East Providence, Rhode Island
  - Teva Investigational Site 10736, Cordova, Tennessee
  - Teva Investigational Site 10701, Franklin, Tennessee
  - Teva Investigational Site 10728, Nashville, Tennessee
  - Teva Investigational Site 10729, Mansfield, Texas
  - Teva Investigational Site 10722, Round Rock, Texas
  - Teva Investigational Site 10699, Salt Lake City, Utah
  - Teva Investigational Site 10700, Roanoke, Virginia

REFERENCES:
- [Result] Wolinsky JS, Borresen TE, Dietrich DW, Wynn D, Sidi Y, Steinerman JR, Knappertz V, Kolodny S; GLACIER Study Group. GLACIER: An open-label, randomized, multicenter study to assess the safety and tolerability of glatiramer acetate 40 mg three-times weekly versus 20 mg daily in patients with relapsing-remitting multiple sclerosis. Mult Scler Relat Disord. 2015 Jul;4(4):370-6. doi: 10.1016/j.msard.2015.06.005. Epub 2015 Jun 14. PMID 26195058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 218 patients with a confirmed and documented RRMS diagnosis were screened for enrollment into this study. Of the 9 patients who were screened but not randomized, 3 were excluded for not meeting the inclusion criteria, 3 were excluded for meeting an exclusion criterion, and 3 were not enrolled for "other" reason.
Groups:
- GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension): Glatiramer acetate (GA) 20 mg in 1 mL SC injection administered every day (QD) for the 4 months of the core period.
  Participants then switched to 40 mg/mL 3 times a week (TIW) dosing if they chose to continue into the extension period.
- GA 40 mg/mL TIW (Core and Extension): Glatiramer acetate (GA) 40 mg in 1 mL SC injection administered three times a week (TIW) for the 4 months of the core period.
  During the Extension period, participants to continue treatment with GA 40 mg/mL TIW until this dose regimen was commercially available for the treatment of RRMS.
Period: Core Period
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Started | 101 | 108
Full Analysis Set | 100 | 108
Completed | 98 | 101
Not Completed | 3 | 7
Not completed — Non-compliance | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4
Period: Extension Period
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Started | 97 (Switchers) | 101 (Non-Switchers)
Full Analysis Set | 95 | 101
Completed | 91 | 97
Not Completed | 6 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension) | Total
Number analyzed (Participants) | 101 | 108 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (9.34) | 50.9 (11.01) | 50.7 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 89 | 172
  Male | 18 | 19 | 37
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 99 | 107 | 206
  Hispanic or Latino | 2 | 0 | 2
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 96 | 100 | 196
  Black | 5 | 5 | 10
  Asian | 0 | 3 | 3
  American Indian or Alaskan Native | 0 | 0 | 0
  Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
Tobacco user [Number; unit: participants]
  Current | 15 | 8 | 23
  Former | 21 | 29 | 50
  Never Smoked | 65 | 71 | 136
Time to First MS Symptom [Mean (Standard Deviation); unit: years] | 16.2 (10.95) | 15.7 (11.10) | 15.9 (11.00)
Time from MS Diagnosis [Mean (Standard Deviation); unit: years] | 12.1 (10.04) | 10.8 (8.55) | 11.5 (9.30)
Number of Relapses in 1 Year Prior to Screening [Mean (Standard Deviation); unit: relapses] | 0.2 (0.41) | 0.2 (0.47) | 0.2 (0.44)
Number of Relapses in 2 Years Prior to Screening [Mean (Standard Deviation); unit: relapses] | 0.4 (0.74) | 0.4 (0.64) | 0.4 (0.69)
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — The Kurtzke Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis. The EDSS quantifies disability in eight Functional Systems (FS):
  * pyramidal
  * cerebellar
  * brainstem
  * sensory
  * bowel and bladder
  * visual
  * cerebral
  * other
  The scale is from 0 (normal neurological examination) to 10 (Death due to MS). A grade of 2.5 refers to a mild disability in one functional system or minimal disability in two functional systems.
  units on a scale | 2.4 (1.38) | 2.5 (1.36) | 2.4 (1.37)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Estimates for Injection-Related Adverse Event Rate Per Year in the Core Period
Description: Injection-related (IR) adverse events refers to all local injection site reactions and/or symptoms or events related to immediate post injection reaction (flushing, chest pain, palpitations, anxiety, dyspnea, throat constriction, and/or urticaria). Rate was calculated as # IR events/the total exposure to study drug in years.
  For cases in which more than 1 IR adverse event started on the same date for the same patient, these were counted as 1 IR adverse event for that patient.
  Parameter statistics were generated from a Poisson regression model with natural log of treatment duration (years) as an offset variable, and adjusted for baseline EDSS score, treatment group, age, sex, number of relapses in the 2 years prior to screening, in which a contrast comparing treatment groups were constructed. Adjusted mean estimates were adjusted estimates of event rates within treatment group.
Time Frame: Day 1 to Month 4
Population: Safety analysis set
Measure: Mean (Standard Error); unit: events per year
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Number analyzed (Participants) | 101 | 108
events per year | 70.403 (11.995) | 35.275 (7.248)
Statistical Analysis 1: Comparison: GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) vs GA 40 mg/mL TIW (Core and Extension); Adjusted mean estimates were adjusted estimates of event rates within treatment group. The treatment effect parameter estimate was a risk ratio of the GA 40 mg/mL TIW treatment group divided by the GA 20 mg/mL QD treatment group. The p value tested whether the risk ratio was significantly different from 1; Test type: Superiority or Other; p = 0.0006, Poisson regression model — The overall significance level for this study was 5% using 2-tailed test; Natural log of treatment duration was an offset variable; adjusted for baseline EDSS, treatment group, age, sex, # relapses 2 years prior to screening; Risk Ratio (RR) = 0.501, 95% CI 2-sided [0.338 to 0.743], Standard Error of Mean 0.101 — GA 40 mg/mL TIW treatment group / GA 20 mg/mL QD treatment group

2. Other Pre Specified Outcome: Percentage of Participants With Adverse Events Other Than Injection Related Reactions During the Core Period and the Extension Period
Description: An adverse event was defined in the protocol as any untoward medical occurrence in a patient that developed or worsened in severity during the conduct of the clinical study of a pharmaceutical product and did not necessarily have a causal relationship to the study drug. This outcome summarizes the % of participants who had AEs other than injection related reactions. Injection-related (IR) adverse events referring to all local injection site reactions and/or symptoms or events related to immediate post injection reaction (flushing, chest pain, palpitations, anxiety, dyspnea, throat constriction, and/or urticaria).
Time Frame: Day 1 to Month 4 (core period); Month 5 to 10 (extension period)
Population: Safety analysis set
Measure: Number; unit: percentage of participants
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Number analyzed (Participants) | 101 | 108
percentage of participants
  Core Period (n=101, 108) | 35.6 | 47.2
  Extension Period (n=97, 101) | 35.1 | 39.6

3. Secondary Outcome: Adjusted Mean Estimates for Injection Site Reaction Event Rate Per Year in the Core Period
Description: This outcome includes injection-related adverse events referring to all local injection site reactions (ISR). Rate was calculated as # ISR events/the total exposure to study drug in years.
  For cases in which more than 1 ISR adverse event started on the same date for the same patient, these were counted as 1 ISR adverse event for that patient.
  Parameter statistics were generated from a Poisson regression model with natural log of treatment duration (years) as an offset variable, and adjusted for baseline EDSS score, treatment group, age, sex, number of relapses in the 2 years prior to screening, in which a contrast comparing treatment groups were constructed. Adjusted mean estimates were adjusted estimates of event rates within treatment group.
Time Frame: Day 1 to Month 4
Population: Safety analysis set
Measure: Mean (Standard Error); unit: events per year
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Number analyzed (Participants) | 101 | 108
events per year | 70.392 (12.007) | 35.200 (7.247)
Statistical Analysis 1: Comparison: GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) vs GA 40 mg/mL TIW (Core and Extension); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0006, Poisson regression model — The overall significance level for this study was 5% using 2-tailed test; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.500, 95% CI 2-sided [0.337 to 0.742], Standard Error of Mean 0.101 — GA 40 mg/mL TIW treatment group / GA 20 mg/mL QD treatment group

4. Secondary Outcome: Change From Baseline to Month 4 in in the Adjusted Mean Participant-Reported Impact on Physical Wellbeing Using Multiple Sclerosis Impact Scale (MSIS-29 PRO) in the Core Period
Description: The physical wellbeing assessment portion of the MSIS-29 is comprised of 20 questions in which participants rate the impact of MS on their day-to-day life during the past two weeks from 1=no impact to 5=extreme impact for a total score of 20-100. Negative change from baseline scores indicate improvement in physical wellbeing over time.
  The estimated change from baseline to month 4 adjusted for months 1 and 2 was generated using a mixed model repeated measures analysis adjusted for baseline MSIS-29 physical score, treatment group, month, treatment by month interaction.
Time Frame: Month 0 (baseline), Months 1, 2, 4 (or early termination visit)
Population: Full analysis set. Some scales/forms were not completed (including partially completed) and therefore not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Number analyzed (Participants) | 85 | 92
units on a scale | 1.536 (0.868) | -0.522 (0.832)
Statistical Analysis 1: Comparison: GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) vs GA 40 mg/mL TIW (Core and Extension); To control for type 1 errors, secondary variables were analyzed only if analysis of the primary variable was statistically significant. Gate-keeping procedures offered further control with this hierarchy: 1. the rate of ISRs 2. change from baseline to month 4 (change - M4) in MSIS-20 physical wellbeing 3. change - M4 in MSIS-20 psychological wellbeing 4. change - M4 in TSQM-9 convenience 5. change - M4 in TSQM-9 overall satisfaction; Test type: Superiority or Other; p = 0.0897, ANCOVA — The overall significance level for this study was 5% using 2-tailed test; In addition to treatment group, month (categorical), treatment-by-month interaction and score at baseline were used as covariates; Mean Difference (Final Values) = -2.058, 95% CI 2-sided [-4.438 to 0.322], Standard Error of Mean 1.206 — GA 40 mg/mL TIW treatment group vs. GA 20 mg/mL QD treatment group

5. Primary Outcome: Injection-Related Adverse Event Rate Per Year in the Extension Period
Description: Injection-related (IR) adverse events refers to all local injection site reactions and/or symptoms or events related to immediate post injection reaction (flushing, chest pain, palpitations, anxiety, dyspnea, throat constriction, and/or urticaria). Rate was calculated as # IR events/the total exposure to study drug in years.
  For cases in which more than 1 IR adverse event started on the same date for the same patient, these were counted as 1 IR adverse event for that patient.
Time Frame: Month 5 up to Month 10
Population: ITT extension analysis set of participants who had at least one injection-related AE
Measure: Number; unit: events per year
Groups:
- Switchers: 40 mg/mL TIW (Extension): Participants who took glatiramer acetate (GA) 20 mg in 1 mL SC injection administered every day (QD) for the 4 months of the core period. Then switched to 40 mg/mL 3 times a week (TIW) dosing in the extension period.
- Non-Switchers: GA 40 mg/mL TIW (Extension): Participants who took glatiramer acetate (GA) 40 mg in 1 mL SC injection administered three times a week in both the core and extension periods.
Arm/Group | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 31 | 33
events per year | 23.1 | 28.0

6. Secondary Outcome: Change From Baseline to Month 4 in in the Adjusted Mean Participant-Reported Impact on Psychological Wellbeing Using Multiple Sclerosis Impact Scale (MSIS-29 PRO) in the Core Period
Description: The psychological wellbeing assessment portion of the MSIS-29 is comprised of 9 questions in which participants rate the impact of MS on their day-to-day life during the past two weeks from 1=no impact to 5=extreme impact for a total score of 9-45. Negative change from baseline scores indicate improvement in psychological wellbeing over time.
  The estimated change from baseline to month 4 adjusted for months 1 and 2 was generated using a mixed model repeated measures analysis adjusted for baseline MSIS-29 psychological score, treatment group, month, treatment by month interaction.
Time Frame: Month 0 (baseline), Months 1, 2 4 (or early termination visit)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Number analyzed (Participants) | 85 | 92
units on a scale | 0.738 (0.533) | 0.016 (0.512)

7. Secondary Outcome: Change From Baseline to Month 4 in in the Adjusted Mean Participant-Reported Treatment Satisfaction Questionnaire for Medication (TSQM-9) Convenience Score in the Core Period
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a psychometric measure of a patient's satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The scores were computed by adding items for each domain, i.e. 1 to 3 for effectiveness, 4 - 6 for convenience and 7 to 9 for global satisfaction. This outcome focuses on convenience items 4-6, with each question graded on a scale of 1 (extreme dissatisfaction) to 7 (extreme satisfaction). TSQM-9 participant perception of convenience score was calculated as: ([sum (Item 4 to Item 6) - 3] divided by 18) * 100. The full range was -100 to 100, with positive change from baseline indicating improvement.
  The estimated change from baseline to month 4 adjusted for months 1 and 2 was generated using a mixed model repeated measures analysis adjusted for baseline TSQM convenience score, treatment group, month, treatment by month interaction.
Time Frame: Month 0 (baseline), Months 1, 2 4 (or early termination visit)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Number analyzed (Participants) | 97 | 105
units on a scale | 1.745 (1.457) | 8.751 (1.399)

8. Secondary Outcome: Change From Baseline to Month 4 in in the Adjusted Mean Participant-Reported Treatment Satisfaction Questionnaire for Medication (TSQM-9) Satisfaction Score in the Core Period
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a psychometric measure of a patient's satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The scores were computed by adding items for each domain, i.e. 1 to 3 for effectiveness, 4 - 6 for convenience and 7 to 9 for global satisfaction. This outcome focuses on global satisfaction, items 7-9. TSQM-9 participant perception of satisfaction score was calculated as: ([sum(Item 7 to Item 9) - 3] divided by 14) * 100. The full range was -100 to 100, with positive change from baseline indicating improvement satisfaction with medication.
  The estimated change from baseline to month 4 adjusted for months 1 and 2 was generated using a mixed model repeated measures analysis adjusted for baseline TSQM convenience score, treatment group, month, treatment by month interaction.
Time Frame: Month 0 (baseline), Months 1, 2 4 (or early termination visit)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | GA 20 mg/mL QD (Core); 40 mg/mL TIW (Extension) | GA 40 mg/mL TIW (Core and Extension)
Number analyzed (Participants) | 97 | 105
units on a scale | 1.555 (1.489) | 0.703 (1.431)

9. Secondary Outcome: Injection Site Reaction Event Rate Per Year in the Extension Period
Description: This outcome includes injection-related adverse events referring to all local injection site reactions (ISR). Rate was calculated as # ISR events/the total exposure to study drug in years.
  For cases in which more than 1 ISR adverse event started on the same date for the same patient, these were counted as 1 ISR adverse event for that patient.
Time Frame: Month 5 up to Month 10
Population: ITT extension analysis set of participants who had injection site reaction AEs.
Measure: Number; unit: events per year
Arm/Group | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 31 | 32
events per year | 22.9 | 28.0

10. Secondary Outcome: Injection Site Reaction Events in the Extension Period
Description: This outcome includes injection-related adverse events referring to all local injection site reactions (ISR).
  For cases in which more than 1 ISR adverse event started on the same date for the same patient, these were counted as 1 ISR adverse event for that patient.
Time Frame: Month 5 up to Month 10
Population: ITT extension analysis set of participants who had injection site reaction AEs.
Measure: Number; unit: events
Arm/Group | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 31 | 32
events | 768 | 976

11. Secondary Outcome: Change From Start of Extension Period (Month 4) to Month 8 (and to Endpoint Visit) in the Participant-Reported Impact on Physical Wellbeing Using Multiple Sclerosis Impact Scale (MSIS-29 PRO)
Description: The physical wellbeing assessment portion of the MSIS-29 is comprised of 20 questions in which participants rate the impact of MS on their day-to-day life during the past two weeks from 1=no impact to 5=extreme impact for a total score of 20-100. Negative change from baseline scores indicate improvement in physical wellbeing.
  The Extension Period endpoint visit was defined as the last observed post-baseline data of the Extension Period.
Time Frame: Month 4 (baseline for extension period), Month 8, endpoint visit
Population: Full analysis set Extension Period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 95 | 101
units on a scale
  Month 8 (n=49, 54) | -0.6 (8.09) | 0.8 (9.53)
  Endpoint visit (n=95, 101) | 1.1 (7.53) | 0.6 (7.60)

12. Secondary Outcome: Change From Start of Extension Period (Month 4) to Month 8 (and to Endpoint Visit) in the Participant-Reported Impact on Psychological Wellbeing Using Multiple Sclerosis Impact Scale (MSIS-29 PRO)
Description: The psychological wellbeing assessment portion of the MSIS-29 is comprised of 9 questions in which participants rate the impact of MS on their day-to-day life during the past two weeks from 1=no impact to 5=extreme impact for a total score of 9-45. Negative change from baseline scores indicate improvement in psychological wellbeing.
  The Extension Period endpoint visit was defined as the last observed post-baseline data of the Extension Period.
Time Frame: Month 4 (baseline for extension period), Month 8, endpoint visit
Population: Full analysis set Extension Period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 95 | 101
units on a scale
  Month 8 (n=49, 54) | 1.2 (4.34) | 0.4 (5.78)
  Endpoint visit (n=95, 101) | 0.9 (5.26) | 0.2 (3.83)

13. Secondary Outcome: Change From Start of Extension Period to Month 8 (and to Endpoint Visit) in in the Participant-Reported Treatment Satisfaction Questionnaire for Medication (TSQM-9) Convenience Score
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a psychometric measure of a patient's satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The scores were computed by adding items for each domain, i.e. 1 to 3 for effectiveness, 4 - 6 for convenience and 7 to 9 for global satisfaction. This outcome focuses on convenience items 4-6, with each question graded on a scale of 1 (extreme dissatisfaction) to 7 (extreme satisfaction). TSQM-9 participant perception of convenience score was calculated as: ([sum (Item 4 to Item 6) - 3] divided by 18) * 100. The full range was -100 to 100, with positive change from baseline indicating improvement.
  The Extension Period endpoint visit was defined as the last observed post-baseline data of the Extension Period.
Time Frame: Month 4 (baseline for extension period), Month 8, endpoint visit
Population: Full analysis set Extension Period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 95 | 101
units on a scale
  Month 8 (n=50, 54) | 4.0 (18.44) | -0.2 (10.41)
  Endpoint visit (n=95, 101) | 4.3 (17.41) | -0.2 (13.10)

14. Primary Outcome: Injection-Related Adverse Events in the Extension Period
Description: Injection-related (IR) adverse events refers to all local injection site reactions and/or symptoms or events related to immediate post injection reaction (flushing, chest pain, palpitations, anxiety, dyspnea, throat constriction, and/or urticaria).
Time Frame: Month 5 up to Month 10
Population: ITT extension analysis set of participants who had at least one injection-related AE
Measure: Number; unit: events
Arm/Group | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 31 | 33
events | 772 | 979

15. Secondary Outcome: Change From Start of Extension Period to Month 8 (and to Endpoint Visit) in in the Participant-Reported Treatment Satisfaction Questionnaire for Medication (TSQM-9) Satisfaction Score
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a psychometric measure of a patient's satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The scores were computed by adding items for each domain, i.e. 1 to 3 for effectiveness, 4 - 6 for convenience and 7 to 9 for global satisfaction. This outcome focuses on global satisfaction, items 7-9. TSQM-9 participant perception of satisfaction score was calculated as: ([sum(Item 7 to Item 9) - 3] divided by 14) * 100. The full range was -100 to 100, with positive change from baseline indicating improvement satisfaction with medication.
  The Extension Period endpoint visit was defined as the last observed post-baseline data of the Extension Period.
Time Frame: Month 4 (baseline for extension period), Month 8, endpoint visit
Population: Full analysis set Extension Period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 95 | 101
units on a scale
  Month 8 (n=50, 54) | -0.3 (14.50) | -1.2 (13.58)
  Endpoint visit (n=95, 101) | -0.0 (14.32) | -1.2 (11.11)

ADVERSE EVENTS:
Time Frame: Day 1 to Month 4 (core period); Month 5 to 10 (extension period)
Groups:
- GA 20 mg/mL QD (Core): Glatiramer acetate (GA) 20 mg in 1 mL SC injection administered every day (QD) for the 4 months of the core period.
- GA 40 mg/mL TIW (Core): Glatiramer acetate (GA) 40 mg in 1 mL SC injection administered three times a week (TIW) for the 4 months of the core period.
Arm/Group | GA 20 mg/mL QD (Core) | GA 40 mg/mL TIW (Core) | Switchers: 40 mg/mL TIW (Extension) | Non-Switchers: GA 40 mg/mL TIW (Extension)
Serious Adverse Events (participants affected / at risk) | 1/101 | 2/108 | 0/97 | 2/101
Other Adverse Events (participants affected / at risk) | 58/101 | 66/108 | 33/97 | 33/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA 20 mg/mL QD (Core) (N=101) | GA 40 mg/mL TIW (Core) (N=108) | Switchers: 40 mg/mL TIW (Extension) (N=97) | Non-Switchers: GA 40 mg/mL TIW (Extension) (N=101)
Ileitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA 20 mg/mL QD (Core) (N=101) | GA 40 mg/mL TIW (Core) (N=108) | Switchers: 40 mg/mL TIW (Extension) (N=97) | Non-Switchers: GA 40 mg/mL TIW (Extension) (N=101)
Injection site bruising (General disorders) | 18 (166) | 8 (8) | 4 (10) | 3 (5)
Injection site erythema (General disorders) | 37 (1331) | 41 (692) | 17 (253) | 21 (436)
Injection site haemorrhage (General disorders) | 11 (43) | 8 (17) | 3 (5) | 7 (10)
Injection site mass (General disorders) | 27 (669) | 28 (381) | 12 (122) | 16 (334)
Injection site pain (General disorders) | 41 (1692) | 42 (803) | 19 (626) | 24 (594)
Injection site pruritus (General disorders) | 15 (398) | 14 (253) | 6 (85) | 8 (81)
Injection site swelling (General disorders) | 24 (594) | 19 (170) | 11 (108) | 7 (89)
Injection site urticaria (General disorders) | 13 (377) | 10 (175) | 4 (77) | 7 (163)
Injection site warmth (General disorders) | 6 (228) | 4 (24) | 2 (27) | 3 (20)
Sinusitis (Infections and infestations) | 3 (3) | 6 (6) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3) | 6 (6) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.